CLINICAL TRIAL: NCT03009721
Title: A Non-interventional, Multi-center, Retrospective Observational Study to Investigate the Effectiveness and Safety of Olostar Tab in Patients With Essential Hypertension and Dyslipidemia (ROSE Study)
Brief Title: Observational Study to Investigate the Effectiveness and Safety of Olostar Tab in Patients With Essential Hypertension and Dyslipidemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DW_DOLO003
Record Dates: First submitted 2017-01-02; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension; Dyslipidemias
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Other: Not applicable-observational study

SUMMARY:
The purpose of this study is to investigate the effectiveness and safety of Olostar Tab in patients with essential hypertension and dyslipidemia

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 19
* Patients have record of blood pressure (SBP/DBP) and LDL-C after prescription of Olostar Tab.

Exclusion Criteria:

* Patients that have participated clinical trials or PMS with Olostar Tab.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with essential hypertension and dyslipidemia
Sampling Method: Probability Sample
Enrollment: 9707 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in blood pressure (SBP/DBP) | At 8 Weeks
Percent change from baseline in LDL-Cholesterol (LDL-C) | At 8 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguk Ilsan University Hospital, Ilsan, South Korea

IPD SHARING:
Plan to Share IPD: No